CLINICAL TRIAL: NCT05330624
Title: Immunogenicity and Safety of Subunit Vaccine of Plague Vaccine (F1+ rV) With Two Immunization Regimens: A Random Phase 2b Clinical Trial
Brief Title: Immunogenicity and Safety of Subunit Vaccine of Plague Vaccine With Two Immunization Regimens
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT083
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Plague
Keywords: Plague vaccine, Immunogenicity, Safety
MeSH Terms: conditions — Plague

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the D0- M1-M6 regimen (Experimental): Adults receive three doses of 1.0 ml plague vaccine at day 0, month 1, and month 6 (referred as the D0-M1-M6 regimen).
  Interventions: Biological: plague vaccine(F1+rV)
- the D0- M2-M6 regimen (Experimental): Adults receive three doses of 1.0 ml plague vaccine at day 0, month 2, and month 6 (referred as the D0-M2-M6 regimen).
  Interventions: Biological: plague vaccine(F1+rV)

INTERVENTIONS:
Biological: plague vaccine(F1+rV) — plague vaccine(F1+rV) (Lanzhou Institute of Biological Products Co.,Ltd) of 1.0ml, three doses

SUMMARY:
Plague is a potentially fatal infection in humans caused by the bacterium Yersinia pestis. Pneumonic plague is typically diagnosed in humans with high mortality. It has a long history for plague as an agent of biowarfare, and pose a serious threat to international security. Althought the killed whole-cell plague vaccine and live attenuated vaccine has been licensed. They are rarely used today because of toxicities, limited evidence for efficacy to prevent plague, and limited commercial availability. In the last twenty years, it have focused on recombinant subunit vaccines which were formed F1 and V antigens as the main composition provide greater protection than vaccines comprised of either subunit alone. This study was aim to exploring the safety and immunogenicity of a new type plague subunit vaccine which comprised natural F1 antigen and recombined V antigen (F1+rV) in two immunization regimens.

DETAILED DESCRIPTION:
Plague is a potentially fatal infection in humans caused by the bacterium Yersinia pestis, transmitted naturally from rodent reservoirs to humans via fleas. Human disease may also result from contact with blood or tissues of infected animals or exposure to aerosolized droplets containing bacteria. Pneumonic plague is typically diagnosed in humans with with high mortality. It has a long history for plague as an agent of biowarfare, and pose a serious threat to international security. In human history, there were three outbreaks of plague all over the world, about 200 million people died from the disease. The increasing trend of plague epidemic in recent years, some regions and countries in the world still has the outbreak of the plague. It implied that safety and safe and effective vaccine is urgently to developing.

Althought the killed whole-cell plague vaccine and live attenuated vaccine has been licensed, these vaccines cause significant adverse reactions, including fever, headache, malaise, lymphadenopathy, erythema and induration at the injection site with high degree of immune variability. They are rarely used today because of toxicities, limited evidence for efficacy to prevent plague, and limited commercial availability. Based on the researches in the last twenty years, it have focused on recombinant subunit vaccines which were formed F1 and V antigens as the main composition provide greater protection than vaccines comprised of either subunit alone. In the primary phase 2a clinical trial, 30μg formulation showed a stronger and sustained immune response. This study was aim to exploring the safety and immunogenicity of a new type plague subunit vaccine which comprised 30μg natural F1 antigen and 30μg recombined V antigen (F1+rV) in two immunization regimens.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-55months old as established by medical history and clinical examination.
* The subjects' guardians are able to understand and sign the informed consent.
* Subjects who can and will comply with the requirements of the protocol.
* Subjects with temperature ≤37.0°C on axillary setting.

Exclusion Criteria:

* Family history of seizures or progressive neurological disease.
* Subject who has a medical history of plague, or had been vaccination of plague vaccine.
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine.
* Any confirmed or suspected autoimmune diseases or immune deficiency disorders, including human immunodeficiency virus (HIV) infection.
* Dysgenopathy or severe chronic disease.
* Pregnant or lactating women, women of reproductive age without contraception.
* Thrombocytopenia or other blood coagulation disorder, taboos of intramuscular injection and collection of blood.
* Difficulty in blood collection.
* Any prior administration of immunodepressant or corticosteroids, and antianaphylactic treatment, cytotoxic therapy in last 6 months.
* Any prior administration of blood products in last 3 month.
* Any prior administration of other research medicines in last 4 weeks.
* Any prior administration of attenuated live vaccine in last 4 weeks.
* Any prior administration of subunit or inactivated vaccines in last 2 weeks.
* Had fever before vaccination, subjects with temperature >37.0°C on axillary setting.
* Any condition that in the opinion of the investigator, may interferes the evaluation of study objectives.

Exclusion Criteria for the other doses:

* Subject who must be excluded according to the exclusion criteria for the first dose
* Grade 3 or above systemic adverse reactions or unacceptable adverse reactions at injection site after the previous inoculation.
* Other reasons in the opinion of the investigator that affect continuing vaccination.

Criteria for postponding of vaccination

-Recovered subject who be sick during the time window of vaccination whether to continue vaccination determined by the investigator according to the requirements of the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 720 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
the GMT of antibodies to F1 antigen on Month 7 post-dose 1 | Month 7 post-dose 1
  the GMT of antibodies to F1 antigen on Month 7 post-dose 1
the GMT of antibodies to rV antigen on Month 7 post-dose 1 | Month 7 post-dose 1
  the GMT of antibodies to rV antigen on Month 7 post-dose 1

SECONDARY OUTCOMES:
The seroconversion of antibodies to F1 antigen on Month 7 post-dose 1 | Month 7 post-dose 1
  The seroconversion of antibodies to F1 antigen on Month 7 post-dose 1
The GMFI of antibodies to F1 antigen on Month 7 post-dose 1 | Month 7 post-dose 1
  The GMFI of antibodies to F1 antigen on Month 7 post-dose 1
The seroconversion of antibodies to rV antigen on Month 7 post-dose 1 | Month 7 post-dose 1
  The seroconversion of antibodies to rV antigen on Month 7 post-dose 1
The GMFI of antibodies to rV antigen on Month 7 post-dose 1 | Month 7 post-dose 1
  the GMFI of antibodies to rV antigen on Month 7 post-dose 1
The GMT of antibodies to F1 antigen on Month 1 post-dose 1 | Month 1 post-dose 1
  The GMT of antibodies to F1 antigen on Month 1 post-dose 1
The GMT of antibodies to rV antigen on Month 1 post-dose 1 | Month 1 post-dose 1
  The GMT of antibodies to rV antigen on Month 1 post-dose 1
The seroconversion of antibodies to F1 antigen on Month1 post-dose 1 | Month 1 post-dose 1
  The seroconversion of antibodies to F1 antigen on Month1 post-dose 1
The seroconversion of antibodies to rV antigen on Month1 post-dose 1 | Month 1 post-dose 1
  The seroconversion of antibodies to rV antigen on Month1 post-dose 1
The GMFI of antibodies to F1 antigen on Month 1 post-dose 1 | Month 1 post-dose 1
  The GMFI of antibodies to F1 antigen on Month 1 post-dose 1
The GMFI of antibodies to rV antigen on Month 1 post-dose 1 | Month 1 post-dose 1
  The GMFI of antibodies to rV antigen on Month 1 post-dose 1
The GMT of antibodies to F1 antigen on Month 2 post-dose 1 | Month 2 post-dose 1
  The GMT of antibodies to F1 antigen on Month 2 post-dose 1
The GMT of antibodies to rV antigen on Month 2 post-dose 1 | Month 2 post-dose 1
  The GMT of antibodies to rV antigen on Month 2 post-dose 1
The seroconversion of antibodies to F1 antigen on Month 2 post-dose 1 | Month 2 post-dose 1
  The seroconversion of antibodies to F1 antigen on Month 2 post-dose 1
The seroconversion of antibodies to rV antigen on Month 2 post-dose 1 | Month 2 post-dose 1
  The seroconversion of antibodies to rV antigen on Month 2 post-dose 1
The GMFI of antibodies to F1 antigen on Month 2 post-dose 1 | Month 2 post-dose 1
  The GMFI of antibodies to F1 antigen on Month 2 post-dose 1
The GMFI of antibodies to rV antigen on Month 2 post-dose 1 | Month 2 post-dose 1
  The GMFI of antibodies to rV antigen on Month 2 post-dose 1
The GMT of antibodies to F1 antigen on Month 3 post-dose 1 | Month 3 post-dose 1
  The GMT of antibodies to F1 antigen on Month 3 post-dose 1
The GMT of antibodies to rV antigen on Month 3 post-dose 1 | Month 3 post-dose 1
  The GMT of antibodies to rV antigen on Month 3 post-dose 1
The seroconversion of antibodies to F1 antigen on Month 3 post-dose 1 | Month 3 post-dose 1
  The seroconversion of antibodies to F1 antigen on Month 3 post-dose 1
The seroconversion of antibodies to rV antigen on Month 3 post-dose 1 | Month 3 post-dose 1
  The seroconversion of antibodies to rV antigen on Month 3 post-dose 1
The GMFI of antibodies to F1 antigen on Month 3 post-dose 1 | Month 3 post-dose 1
  The GMFI of antibodies to F1 antigen on Month 3 post-dose 1
The GMFI of antibodies to rV antigen on Month 3 post-dose 1 | Month 3 post-dose 1
  The GMFI of antibodies to rV antigen on Month 3 post-dose 1
The GMT of antibodies to F1 antigen on Month 6 post-dose 1 | Month 6 post-dose 1
  The GMT of antibodies to F1 antigen on Month 6 post-dose 1
The GMT of antibodies to rV antigen on Month 6 post-dose 1 | Month 6 post-dose 1
  The GMT of antibodies to rV antigen on Month 6 post-dose 1
The seroconversion of antibodies to F1 antigen on Month 6 post-dose 1 | Month 6 post-dose 1
  The seroconversion of antibodies to F1 antigen on Month 6 post-dose 1
The seroconversion of antibodies to rV antigen on Month 6 post-dose 1 | Month 6 post-dose 1
  The seroconversion of antibodies to rV antigen on Month 6 post-dose 1
The GMFI of antibodies to F1 antigen on Month 6 post-dose 1 | Month 6 post-dose 1
  The GMFI of antibodies to F1 antigen on Month 6 post-dose 1
The GMFI of antibodies to rV antigen on Month 6 post-dose 1 | Month 6 post-dose 1
  The GMFI of antibodies to rV antigen on Month 6 post-dose 1
The GMT of antibodies to F1 antigen on Month 9 post-dose 1 | Month 9 post-dose 1
  The GMT of antibodies to F1 antigen on Month 9 post-dose 1
The GMT of antibodies to rV antigen on Month 9 post-dose 1 | Month 9 post-dose 1
  The GMT of antibodies to rV antigen on Month 9 post-dose 1
The seroconversion of antibodies to F1 antigen on Month 9 post-dose 1 | Month 9 post-dose 1
  The seroconversion of antibodies to F1 antigen on Month 9 post-dose 1
The seroconversion of antibodies to rV antigen on Month 9 post-dose 1 | Month 9 post-dose 1
  The seroconversion of antibodies to rV antigen on Month 9 post-dose 1
The GMFI of antibodies to F1 antigen on Month 9 post-dose 1 | Month 9 post-dose 1
  The GMFI of antibodies to F1 antigen on Month 9 post-dose 1
The GMFI of antibodies to rV antigen on Month 9 post-dose 1 | Month 9 post-dose 1
  The GMFI of antibodies to rV antigen on Month 9 post-dose 1
The GMT of antibodies to F1 antigen on Month12 post-dose 1 | Month 12 post-dose 1
  The GMT of antibodies to F1 antigen on Month12 post-dose 1
The GMT of antibodies to rV antigen on Month12 post-dose 1 | Month 12 post-dose 1
  The GMT of antibodies to rV antigen on Month12 post-dose 1
The seroconversion of antibodies to F1 antigen on Month 12 post-dose 1 | Month 12 post-dose 1
  The seroconversion of antibodies to F1 antigen on Month 12 post-dose 1
The seroconversion of antibodies to rV antigen on Month 12 post-dose 1 | Month 12 post-dose 1
  The seroconversion of antibodies to rV antigen on Month 12 post-dose 1
The GMFI of antibodies to F1 antigen on Month 12 post-dose 1 | Month 12 post-dose 1
  The GMFI of antibodies to F1 antigen on Month 12 post-dose 1
The GMFI of antibodies to rV antigen on Month 12 post-dose 1 | Month 12 post-dose 1
  The GMFI of antibodies to rV antigen on Month 12 post-dose 1
The GMT of antibodies to F1 antigen on Month18 post-dose 1 | Month 18 post-dose 1
  The GMT of antibodies to F1 antigen on Month18 post-dose 1
The GMT of antibodies to rV antigen on Month18 post-dose 1 | Month 18 post-dose 1
  The GMT of antibodies to rV antigen on Month18 post-dose 1
The seroconversion of antibodies to F1 antigen on Month 18 post-dose 1 | Month 18 post-dose 1
  The seroconversion of antibodies to F1 antigen on Month 18 post-dose 1
The seroconversion of antibodies to rV antigen on Month 18 post-dose 1 | Month 18 post-dose 1
  The seroconversion of antibodies to rV antigen on Month 18 post-dose 1
The GMFI of antibodies to F1 antigen on Month 18 post-dose 1 | Month 18 post-dose 1
  The GMFI of antibodies to F1 antigen on Month 18 post-dose 1
The GMFI of antibodies to rV antigen on Month 18 post-dose 1 | Month 18 post-dose 1
  The GMFI of antibodies to rV antigen on Month 18 post-dose 1
The GMT of antibodies to F1 antigen on Month24 post-dose 1 | Month 24 post-dose 1
  The GMT of antibodies to F1 antigen on Month24 post-dose 1
The GMT of antibodies to rV antigen on Month24 post-dose 1 | Month 24 post-dose 1
  The GMT of antibodies to rV antigen on Month24 post-dose 1
The seroconversion of antibodies to F1 antigen on Month 24 post-dose 1 | Month 24 post-dose 1
  The seroconversion of antibodies to F1 antigen on Month 24 post-dose 1
The seroconversion of antibodies to rV antigen on Month 24 post-dose 1 | Month 24 post-dose 1
  The seroconversion of antibodies to rV antigen on Month 24 post-dose 1
The GMFI of antibodies to F1 antigen on Month 24 post-dose 1 | Month 24 post-dose 1
  The GMFI of antibodies to F1 antigen on Month 24 post-dose 1
The GMFI of antibodies to rV antigen on Month 24 post-dose 1 | Month 24 post-dose 1
  The GMFI of antibodies to rV antigen on Month 24 post-dose 1
Proportion of subjects reporting adverse events | Day 30 post-each dose
  Proportion of subjects reporting adverse events within 30 days post-each dose
Proportion of subjects with serious adverse events (SAE)occurring throughout the trial | Day 0 up to month 12 post dose 1
  Proportion of subjects with serious adverse events (SAE)occurring throughout the trial from day 0 to month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Master, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China